CLINICAL TRIAL: NCT00002056
Title: A Controlled Trial Comparing the Efficacy of Aerosolized Pentamidine and Parenteral / Oral Trimethoprim - Sulfamethoxazole in the Treatment of Pneumocystis Carinii Pneumonia in AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LyphoMed (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 023A; 87-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-08

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Injections, Intravenous; Administration, Oral; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
This is a randomized double-blinded controlled study comparing aerosolized pentamidine with trimethoprim plus sulfamethoxazole (TMP / PurposeX). The latter drug will be administered intravenously for at least 5 days, then changed to oral administration if warranted by the patient's clinical condition.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine as long as such therapy is suspended prior to randomization and not reinstituted until therapy for the acute episode is completed.

Pneumocystis carinii pneumonia (PCP) in an adult who is HIV positive by ELISA, HIV culture, or p24 antigenemia, or is a member of a risk group for HIV infection (homosexual or bisexual men, intravenous drug abusers, recipients of HIV infected blood products, and the sexual partners of the foregoing groups).

* The patient must have a resting Alveolar - arterial oxygen (A-a) DO2 less than 30 mmHg on room air at all ACTG sites, except San Francisco General Hospital. Other sites will enter patients up to a resting (A-a) DO2 = or < 55 mmHg on room air.

Prior Medication:

Allowed:

* Zidovudine as long as such therapy is suspended prior to randomization and not reinstituted until therapy for the acute episode is completed.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Dyspnea.
* Cough.
* Bronchospasm.
* History of a major adverse reaction to pentamidine or sulfonamide containing preparations.

Patients with the following will be excluded:

* Inability to cooperate with aerosol administration because of dyspnea, cough, bronchospasm, or other reasons.
* History of a major adverse reaction to pentamidine or sulfonamide containing preparations.
* In the opinion of the investigator, the patient would not complete therapy or follow-up for social reasons.

Prior Medication:

Excluded within 14 days of study entry:

* Systemic steroids above adrenal replacement doses.
* Excluded within 6 weeks of study entry:
* Other antiprotozoal regimen for this episode such as trimethoprim / sulfamethoxazole (TMP / PurposeX).
* Pyrimethamine.
* Fansidar.
* Pentamidine.
* Eflornithine (DFMO).
* Dapsone, whether therapeutic or prophylactic, or any of these agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- LyphoMed Inc, Rosemont, Illinois, United States

REFERENCES:
- [Background] Montgomery AB, Edison RE, Sattler F, Hopewell P, Mason G, Feigal DW. Aerosolized pentamidine vs. trimethoprim/sulfamethoxazole for acute Pneumcoystis carinii pneumonia (PCP): a randomized double blind trial. Int Conf AIDS. 1990 Jun 20-23;6(1):220 (abstract no ThB395)